CLINICAL TRIAL: NCT01729884
Title: Phase II Study to Evaluate the Development of HER2/Neu (HER2)-Specific Memory T Cells After HER2 Peptide-based Vaccination in Patients With Advanced Stage Her2+ Breast Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Hormone Receptor Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ended early due to slow enrollment
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7905; NCI-2012-02223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7905 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P50CA138293 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (HER-2/neu peptide vaccine) (Experimental): Patients receive HER-2/neu peptide vaccine ID once monthly for 3 months.
  Interventions: Biological: HER-2/neu peptide vaccine

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine — Given ID
  Other Names: HER-2

SUMMARY:
This phase II trial studies how well vaccine therapy works in treating patients with stage IV hormone receptor positive breast cancer. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantify and characterize human epidermal growth factor receptor 2 (HER2)-specific central memory T cell (TCM) and effector memory T cell (TEM) subsets in peripheral blood mononuclear cell (PBMC) of patients vaccinated with a HER2 cytotoxic T lymphocyte (CTL) peptide-based vaccine.

II. To evaluate the feasibility of expanding HER2-specific effector T cells (TE) derived from HER2-specific TCM or TEM precursors in patients vaccinated with a HER2 CTL peptide-based vaccine and characterize their function.

SECONDARY OBJECTIVES:

I. To evaluate the safety of administering a HER2 CTL peptide-based vaccine in patients who are receiving trastuzumab and/or lapatinib (lapatinib ditosylate).

OUTLINE:

Patients receive HER-2/neu peptide vaccine intradermally (ID) once monthly for 3 months.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2+ stage IV breast cancer that have been maximally treated and not in a complete remission
* Patients must have measurable disease per imaging studies performed within 60 days of enrollment as described below:

  * Extra skeletal disease that can be measured with conventional or spiral computed tomography (CT) techniques
  * Skeletal or bone-only disease that is measurable by fludeoxyglucose F 18 (FDG) positron emission tomography (PET) or magnetic resonance imaging (MRI)
* Patients can be receiving trastuzumab and/or lapatinib and/or hormonal therapy and/or bisphosphonate therapy
* HER2 overexpression in the primary tumor or metastasis by immunohistochemistry (IHC) of 3+, or documented gene amplification by fluorescent in situ hybridization (FISH) analysis
* Patients must be human leukocyte antigen (HLA)-A2 positive
* Eastern Cooperative Oncology Group (ECOG)/Zubrod scale of =< 1
* Patients must be off immunosuppressive treatments (i.e., chemotherapy or systemic steroids) 3 weeks prior to first vaccine
* Patients on trastuzumab must have a baseline left ventricular ejection fraction (LVEF) measured by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) >= the lower limit of normal for the facility within 3 months of enrollment to study
* Subjects of reproductive ability must agree to use contraceptives during the entire study period

Exclusion Criteria:

* White blood cell (WBC) < 3000/mm^3
* Hemoglobin (Hgb) < 10 mg/dl
* Platelets < 100,000/mm^3
* Serum creatinine > 2.0 mg/dl
* Serum bilirubin > 1.5 x upper limit of normal
* Any contraindication to receiving sargramostim (GM-CSF) based vaccine products
* Concurrent enrollment in other treatment studies
* New York Heart Association functional class III-IV heart failure, symptomatic pericardial effusion, or unstable angina
* Pregnant or breast-feeding women
* History of disorders associated with immunosuppression such as human immunodeficiency virus (HIV)
* Active brain metastasis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quantification and characterization of HER2-specific TCM and TEM subsets in PBMC | Up to 4 weeks
  Wilson score 90% confidence intervals will be reported.
Evaluation of function and phenotype of HER2-specific TE cells derived from HER2-specific TCM and TEM subsets | Up to 4 weeks
  Wilson score 90% confidence intervals will be reported. Determined by flow cytometry and reported using descriptive statistics and graphical summaries.

SECONDARY OUTCOMES:
The number of subjects reporting adverse events, evaluated according to the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4 weeks
  All, severe or worse, serious and related events will be quantified.
The percent of subjects recording adverse events, evaluated according to the CTEP CTCAE version 4.0 | Up to 4 weeks
  All, severe or worse, serious and related events will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States